CLINICAL TRIAL: NCT04670965
Title: Release Kinetics of rhBMP-2 Using E-PRF as an Autologous Carrier: An in Vitro Analysis
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Maria L. Geisinger, DDS, MS, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300005939; UAB-Perio (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Bone Loss
Keywords: Platelet concentrates; Platelet-rich fibrin; Growth factor; Bone morphogenic protein
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood will be harvested to form L-PRF membranes, which will be used in in vitro clinical assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- E-PRF/rhBMP-2 (similar ratios): Subjects will be used to procure the venous blood samples to make the enhanced platelet rich fibrin (E-PRF). Subjects have an established treatment plan that utilizes autologous PRF as an adjunctive biologic therapy during periodontal treatment.
  Interventions: Biological: E-PRF/rhBMP-2 (similar ratios)
- E-PRF/ACS/rhBMP-2: Subjects will be used to procure the venous blood samples to make the enhanced platelet rich fibrin (E-PRF). Subjects have an established treatment plan that utilizes autologous PRF as an adjunctive biologic therapy during periodontal treatment.
  Interventions: Biological: E-PRF/ACS/rhBMP-2
- rhBMP-2/E-PRF: Subjects will be used to procure the venous blood samples to make the enhanced platelet rich fibrin (E-PRF). Subjects have an established treatment plan that utilizes autologous PRF as an adjunctive biologic therapy during periodontal treatment.
  Interventions: Biological: rhBMP-2/E-PRF
- E-PRF only: Subjects will be used to procure the venous blood samples to make the enhanced platelet rich fibrin (E-PRF). Subjects have an established treatment plan that utilizes autologous PRF as an adjunctive biologic therapy during periodontal treatment.
  Interventions: Biological: E-PRF only

INTERVENTIONS:
Biological: E-PRF/rhBMP-2 (similar ratios) — During its preparation, 1.5 mg/ml rhBMP-2 will be incorporated into standardized samples to assure similar E-PRF to rhBMP-2 ratios. To allow for consistency across all samples, standardized E-PRF volume will be established using formation templates. Following its preparation, the E-PRF/rhBMP2 scaffold will undergo a standard in vitro assay to investigate growth factor release over time (ELISA quantification assay). Briefly, the e-PRF/rhBMP2 scaffold will be placed in a shaking incubator at 37 degree Celsius and assessed for growth factor release of rhBMP-2 over time.
  Groups: E-PRF/rhBMP-2 (similar ratios)
Biological: E-PRF/ACS/rhBMP-2 — rhBMP-2 diluted to account for the additional volume from the E-PRF in other samples will be loaded onto lyophilized absorbable collagen sponges as per the package insert. After the addition of the rhBMP-2, the ACS will be cut into 2mm x 2mm pieces and incorporated into the E-PRF membrane. Following its preparation, rhBMP-2 release from the E-PRF/ACS/rhBMP2 scaffold will be quantified using the ELISA quantification assay as described above.
  Groups: E-PRF/ACS/rhBMP-2
Biological: rhBMP-2/E-PRF — rhBMP-2 diluted to account for the additional volume from the E-PRF in other samples will be loaded onto lyophilized absorbable collagen sponges as per the package insert. Rh-BMP2 release will be quantified using the ELISA quantification assay as described above
  Groups: rhBMP-2/E-PRF
Biological: E-PRF only — E-PRF will be prepared and standardized, but no rhBMP-2 will be added to the material. After preparation, the E-PRF scaffold assayed via ELISA quantification assay as described above to determine the release (if any) of intrinsic BMP-2 from the platelet concentrate scaffold.
  Groups: E-PRF only

SUMMARY:
This study is seeking to evaluate the binding of a commercially-available, recombinant human osteoinductive growth factor, rhBMP-2, to a human blood derived product scaffold, enhanced Platelet-rich fibrin (E-PRF), and the release of such a growth factor over time in an in vitro (laboratory) environment. The investigators will compare these release kinetics to those of the FDA approved carrier for rhBMP-2, an absorbable collagen sponge (ACS), a combination of E-PRF and ACS, and E-PRF alone.

DETAILED DESCRIPTION:
Innovations in biomedicine and recombinant protein technology show promising advances for the regeneration of advanced alveolar defects. Recombinant growth factors and biologics encourage minimally invasive procedures with improved clinical outcomes/healing times in complex oral surgery procedures. Recombinant human bone morphogenic protein-2 (rhBMP-2) is a morphogen that is a well-known regulator of bone formation1 and has been widely studied for bone reconstructive treatments.2-6 RhBMP-2 is currently commercially available and loaded on an absorbable collagen sponge (ACS). This recombinant growth factor has been approved by the US Food and Drug Administration as an alternative to autogenous bone grafting in sinus augmentation and localized alveolar ridge augmentation for defects associated with extraction sockets. It is also used off-label for vertical bone augmentation. However, there are limitations of the ACS as a carrier because it is compressible and does not ideally support soft tissues to maintain space for osteogenesis to occur. Furthermore, the release kinetics of rhBMP-2 in a standardized in vitro environment from its ACS carrier are unknown and it is further unknown how such release would compare to the use of other carriers. Subcutaneous implantation in rats and implantation at orthotropic sites in rats and rabbits has also revealed that rhBMP-2-loaded ACS has a release of rhBMP-2 over 21 days with a half-life of 2 days. The use of an alternative delivery system may retain and sequester rhBMPs at the target site and extend its growth factor release over time. This may be clinically relevant as prolonging tissue exposure to an osteoinductive growth factor like rhBMP-2 could extend the period of osteoblastic bone deposition and improve repair at regenerative sites. E-PRF as an autologous carrier for rhBMP-2 may be advantageous based on its resorption properties of up to 4-6 months, as well as its ability to support the healing process due to the slow and gradual release of several growth factors including, PDGF-AA, PDGF-BB, TGF- β1,VEGF, IGF, and EGF. This study aims to quantify the release of rhBMP-2 over a 120 day period with the use of a novel delivery system, E-PRF.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* At least 18 years old
* Must be a patient of the UAB Dental School
* Able to read and understand informed consent document
* Previously treatment planned for a periodontal procedure that will utilize PRF, i.e. requiring venipuncture, as a part of the routine clinical care.

Exclusion Criteria:

* Non-English speaking
* Less than 18 years old
* Smokers/tobacco users (>10 cigarettes/day)
* Patients with systemic pathologies or conditions contraindicating oral surgical procedures or adversely affecting wound healing as assessed by Board Certified Periodontal faculty at UAB Department of Periodontology
* Patient-reported serious adverse events reported with venipuncture, blood sample collection, and/or blood donation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants must be at least 18 years old with demonstrated ability to understand and consent to the proposed study procedures. Subjects treated in the UAB School of Dentistry Periodontal Clinic and scheduled for procedures using platelet rich fibrin (PRF) were performed.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
To quantify any difference between test groups in the release of rhBMP-2 after application to E-PRF and ACS, E-PRF, and ACS. | From baseline to 6 months
  The quanitites of rhBMP-2 at all time points from all groups will be compared using statistical analysis by two-way ANOVA with Bonferroni test.

SECONDARY OUTCOMES:
To more assess the capability of E-PRF without added rhBMP-2 to release any intrinsic autologous BMP-2 under experimental conditions. | From baseline to 6 months
  The quanitites of rhBMP-2 at all time points from all groups will be compared using statistical analysis by two-way ANOVA with Bonferroni test.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Geisinger, DDS, MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States